CLINICAL TRIAL: NCT03490864
Title: Strengthening Circadian Signals to Enhance Cardiometabolic Functions
Brief Title: Strengthening Circadian Signals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Phyllis Zee, Professor of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU00206038
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Improving Cardiometabolic Outcomes in Adults
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomized controlled trial where each participant will receive one of four intervention types. Subjects will be randomized at baseline visit to one of four arms using a randomized block design to achieve balanced groups. Randomization will be stratified by sex. The allocation will be created using an online randomization tool. This study will include a 6 week four arm field intervention to evaluate the independent effect of meal of timing or melatonin as well as their combined effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Meal timing + Melatonin (Experimental): This arm will consist of imposing a minimum overnight fasting period of 12 hours and a maximum of 16 hours (with exception of water and other non-caloric beverages), beginning 3 hours before their habitual bed time. This arm will also include a 1mg melatonin supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Melatonin 1 mg; Other: Meal Timing
- Meal timing + Placebo (Experimental): This arm will consist of imposing a minimum overnight fasting period of 12 hours and a maximum of 16 hours (with exception of water and other non-caloric beverages), beginning 3 hours before their habitual bed time. This arm will also include a melatonin placebo (lactose) supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Placebos; Other: Meal Timing
- Melatonin (Experimental): This arm will continue to eat at their habitual meal times, and maintain their average habitual caloric and macronutrient intake. No extended overnight fasting will be imposed. This arm will include a 1mg melatonin supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Melatonin 1 mg; Other: NON Meal Timing
- Placebo (Placebo Comparator): This arm will continue to eat at their habitual meal times, and maintain their average habitual caloric and macronutrient intake. No extended overnight fasting will be imposed. This arm will also include a melatonin placebo (lactose) supplementation given daily during the intervention
  Interventions: Dietary Supplement: Placebos; Other: NON Meal Timing

INTERVENTIONS:
Dietary Supplement: Melatonin 1 mg — Melatonin (1mg) or placebo will be administered daily during the intervention. Melatonin capsules will be obtained from Life Extension (Ft. Lauderdale, FL). The investigational drug pharmacy (IDP) at Northwestern Memorial Hospital will encapsulate the melatonin pills so the placebo (lactose) and melatonin pills appear identical. We have worked with this IDP on other projects. The investigators on this study have experience in administering melatonin for investigational and clinical purposes.
  Arms: Meal timing + Melatonin; Melatonin
Dietary Supplement: Placebos — Melatonin (1mg) or placebo will be administered daily during the intervention. Melatonin capsules will be obtained from Life Extension (Ft. Lauderdale, FL). The investigational drug pharmacy (IDP) at Northwestern Memorial Hospital will encapsulate the melatonin pills so the placebo (lactose) and melatonin pills appear identical. We have worked with this IDP on other projects. The investigators on this study have experience in administering melatonin for investigational and clinical purposes.
  Arms: Meal timing + Placebo; Placebo
Other: Meal Timing — Subjects are instructed to maintain an extended overnight fasting period of 12-16 hours.
  Other Names: Extended overnight fasting (EOF)
  Arms: Meal timing + Melatonin; Meal timing + Placebo
Other: NON Meal Timing — Subjects are instructed to maintain their habitual meal timing.
  Other Names: NON Extended overnight fasting (nEOF)
  Arms: Melatonin; Placebo

SUMMARY:
There is a growing body of evidence from both laboratory and field studies that disrupted circadian function, particularly decreased amplitude and stability of rhythmic behaviors represent significant risk factors for cardiometabolic disease (CMD) in humans. The exciting evidence of the ubiquity of circadian clocks in all tissues and their critical role in metabolism, not only opens up new avenues for understanding the mechanistic interactions between central and peripheral clocks in cardiometabolic disease pathogenesis, but also to develop therapeutic interventions to re-establish synchrony between central and peripheral clocks with each other and with the external physical and social environments. Feeding has been shown to synchronize clocks in peripheral tissues. Animal studies have demonstrated that restricting feeding to the active period decreases CMD risk, while in humans decreased caloric intake in the evening is associated with a lower body mass index (BMI). The amplitude of melatonin can be considered a marker of robustness of central circadian function, but melatonin also has physiological effects beyond circadian regulation throughout the body. Recent observations have demonstrated that having a low melatonin level is a risk factor for incident diabetes and hypertension independent of sleep duration. Together, the evidence suggests that strategies aimed at synchronizing feeding behavior and enhancing the nocturnal melatonin signal can positively impact cardiometabolic function.

We propose to take an innovative approach that combines the recent data on the role of feed/fast patterns on clock regulated metabolic activity and the reemergence of scientific interest of the central and peripheral effects of melatonin on cardiometabolic function to elucidate the physiological and molecular mechanisms that underlie the relationship between circadian dysregulation and obesity associated CMD risk. This will be accomplished by strengthening the amplitude of circadian metabolic signals via meal timing and enhancement of nocturnal circadian signaling with exogenous melatonin in overweight and obese middle aged and older adults. In addition, this study will provide crucial information regarding the importance of circadian timing for the design of future clinical trials on CMD in overweight and obese adults. This is a critical time in the lifespan when circadian based strategies for prevention and treatment are most likely to have the greatest impact on CMD risk. This project will enroll 100 adults (40-54 years) to participate in a parallel (4 arm intervention) placebo controlled study to determine whether a six- week program of meal timing and/or low dose (1 mg) melatonin administration will enhance circadian amplitude and enhance cardiometabolic function, as well as to evaluate the potential beneficial effects of a regimen that combines both approaches. The results from this study will demonstrate novel mechanistically based approaches for maintaining and improving circadian-metabolic health during a critical time in the lifespan when there is a rapid increase in the prevalence of CMD.

ELIGIBILITY:
Inclusion Criteria:

* Adults 35-54 years old.
* BMI ≥25 to <45
* Regular eating schedule

  * consuming at least 2 meals/day
* Regular sleep schedules (deviation ≤2 hours in daily mid-sleep time)

  * self-reported average sleep duration of ≥6.5 hours,
  * habitual mid-sleep time 2-5am,
  * habitual time in bed of ≤ 9 hours,
* Habitual overnight fast of ≤ 13 hour

  * Determined by a mean overnight fast ≤ 13 hours over 3 days of self-monitoring of food intake at screening
* HbA1C<6.5

Exclusion Criteria:

* History or current diagnosis of a primary sleep disorder (Chronic insomnia, restless leg syndrome, parasomnias, sleep apnea)
* AHI ≥30
* Current anemia
* Diagnosis of diabetes or currently on any medications for diabetes.
* Endocrine dysfunction including PCOS
* History of cognitive or other neurological disorders
* History of DSM-V criteria for any major psychiatric disorder
* Night Eating Syndrome (NES)
* Beck depression Index (BDI) of ≥16 indicating moderate depression
* Mini mental status Exam <26 indicating cognitive impairment.
* Unstable or serious medical conditions
* Individuals with pacemakers, defibrillators, mediation pumps, or any other implanted device.
* Any GI disease that requires dietary adjustment
* Current or use within last month of melatonin
* Current use of psychoactive, hypnotic, stimulants, or pain medications.
* Current use of hormone replacement therapy
* Shift work or other self-imposed irregular sleep schedules.
* History of habitual smoking (≥6 cigarettes/week)
* Caffeine consumption >400 mg/day
* Medically managed or self-reported weight loss program within past 6 months
* Bariatric weight loss surgery.
* Blindness or visual impairment other than glasses
* Allergic to heparin.
* Adults unable to consent will be excluded.
* Pregnant women will be excluded.
* Prisoners will be excluded.
* Individuals who are not yet adults (infants, children, teenagers) will be excluded.

Ages: 35 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Matsuda Index | 8 Weeks
  The matsuda index of whole body index sensitivity will be calculated to explore the effect of sleep and circadian rhythms on the relationship between EOF, Melatonin, and CMD.
Nocturnal Blood Pressure Dipping | 8 Weeks
  Defined as a ratio of sleep Blood Pressure to wake Blood Pressure <0.90.
Melatonin Amplitude | 8 Weeks.
  The melatonin amplitude will be calculated to determine the effects of interventions on sleep and CMD outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Zee, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided